CLINICAL TRIAL: NCT02460874
Title: A Pilot Study and Phase II Double Blind Placebo Controlled Randomized Trial Examining the Safety and Efficacy of Glyburide as Prophylaxis Against Cerebral Edema in Patients Receiving Radiosurgery for Brain Metastases
Brief Title: Glyburide vs Placebo as Prophylaxis Against Cerebral Edema in Patients Receiving Radiosurgery for Brain Metastases (RAD 1502/UAB 1593)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Drexell Hunter Boggs, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-16063003
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Edema; Brain Metastases
Keywords: Brain Metastases; Stereotactic Radiosurgery; Glyburide
MeSH Terms: conditions — Brain Edema; Brain Neoplasms | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pilot Portion (Experimental): Step 1: Patients with brain metastases requiring SRS and not taking corticosteroids 5 days prior to SRS. Treatment planning MRI may be done within 21 days prior to SRS treatment.
  Step 2: Take Glyburide 1.25mg (twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education- begin glucose monitoring (4 times a day).
  Step 3: 1 week after SRS, return to clinic to review glucose logs- continue glyburide and blood glucose monitoring.
  Step 4: 1 month after SRS, discontinue both glyburide and blood glucose monitoring, undergo MRI.
  Step 5: 3 months after SRS, undergo MRI.
  Interventions: Drug: Glyburide
- Randomized Portion (Placebo Comparator): Step 1: Patients with brain metastases requiring SRS and not taking corticosteroids 5 days prior to SRS.Treatment planning MRI may be done within 21 days prior to SRS treatment.
  Step 2: Randomization (1:1)
  * Group 1: take Glyburide (1.25mg, twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education. Begin glucose monitoring (once a day) {This portion will be double blinded}.
  * Group 2: Take Placebo (1 pill, twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education. Begin glucose monitoring (once a day) {This portion will be double blinded}.
  Step 3: 1 week after SRS, return to clinic to review glucose logs, continue investigation medication, but discontinue glucose monitoring.
  Step 4: 1 month after SRS, discontinue investigation medication, undergo MRI.
  Step 5: 3 months after SRS, undergo MRI.
  Interventions: Drug: Glyburide; Other: Placebo

INTERVENTIONS:
Drug: Glyburide — 1.25mg, twice a day
Other: Placebo — 1.25mg, twice a day
  Arms: Randomized Portion

SUMMARY:
Primary Objectives:

Pilot Portion: To determine the feasibility and safety of administering oral glyburide to non-diabetic patients receiving stereotactic radiosurgery (SRS) for newly diagnosed brain metastases.

Randomized Portion: To determine the number of patients with newly diagnosed brain metastases who have an increase in edema as measured on volumetric FLAIR imaging and the number of patients that require dexamethasone administration (or any corticosteroid administration with the purpose of treating cerebral edema) from the day of SRS to one month follow-up MRI in the group receiving glyburide versus placebo.

DETAILED DESCRIPTION:
Many patients with cancer that has spread to the brain have side effects caused by swelling around the tumors. A common treatment for this swelling is a medicine called dexamethasone. Dexamethasone is a steroid. Long-term use of steroids has several known side effects.

Recent studies have shown that a drug commonly used in to control high blood sugar in diabetes, called glyburide, can decrease brain swelling in patients with brain damage or stroke. Animal studies have shown that this drug may also reduce swelling from tumors in the brain. Researchers are interested in whether glyburide could treat brain swelling as well as dexamethasone with fewer side effects.

This study is being done to see whether glyburide is safe to be used in patients without diabetes in combination with receiving SRS for brain metastases. This study will also find out if glyburide will decrease brain swelling in patients that get radiosurgery (SRS) for brain metastases. This study will also find out if taking glyburide will decrease the chance of needing steroids due to brain swelling that is causing symptoms. It is not yet known, but it is the investigators' hope that glyburide will both decrease brain swelling and lessen the chance of needing steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed brain metastases deemed to be eligible for radiosurgery.
* Subject must have cytologically or histologically confirmed malignancy (this is the original malignancy, not the brain metastases).
* A diagnostic contrast-enhanced MRI of the brain must be performed within 60 days prior to registration. The contrast-enhancing intraparenchymal brain tumor must be well visualized.
* History and physical with neurological examination, height, and weight within 14 days prior to registration
* No dexamethasone use (or any other corticosteroid use with the purpose of treating cerebral edema) starting 5 days prior to SRS. Patients may be tapered to meet this criterion if deemed safe by the treating physician.
* Women of child-bearing potential (e.g. not post-menopausal or permanently sterilized women) must have a negative pregnancy test obtained within 14 days prior to registration. This is to prevent potential harm to the fetus by glyburide and radiotherapy.
* CBC with differential and CMP including Liver Function Tests (LFTs) obtained within 14 days prior to registration and meeting the following requirements:

  * Creatinine Clearance ≥ 50 mL/min.
  * Total Bilirubin < 1.5 x the upper limit of normal (ULN).
  * ALT and AST ≤ 2.5 x ULN.
  * Glucose ≥ 80 mg/dL.
  * Hemoglobin ≥ 7 mg/dL.
  * Absolute Neutrophil Count > 100 cells/mm3.
* For the Randomized Portion only: Subject must have at least 2 of the following risk factors: {For the Pilot Portion, it is not required that patients have the risk factors mentioned in Inclusion Criteria 9.}

  * Pretreatment Edema/Tumor ratio (≥ 35:1) as contoured on a baseline MRI obtained at most 60 days prior to registration. Patients are allowed to have Whole Brain Radiotherapy (WBRT) or corticosteroid use between the time of pretreatment MRI and SRS (as long as the corticosteroids can be safely tapered at least 5 days prior to the treatment planning MRI and WBRT is at least 4 days prior to registration).
  * Greater than 40 pack year history of smoking cigarettes.
  * Whole Brain Radiotherapy at least 4 days and no more than 1 year prior to registration.
  * RPA Class III.

Exclusion Criteria:

* Known sulfonylurea treatment within 7 days prior to registration. Sulfonylureas include glyburide/glibenclamide (Diabeta, Glynase); glyburide plus metformin (Glucovance); glimepiride (Amaryl); repaglinide (Prandin); nateglinide (Starlix); glipizide (Glucotrol, GlibeneseR, MinodiabR); gliclazide (DiamicronR); tolbutamide (Orinase, Tolinase); and glibornuride (Glutril).
* Diffuse Leptomeningeal metastases.
* Known allergy to sulfa or specific allergy to sulfonylurea drugs.
* Use of VEGF inhibitors within 10 days prior to registration.
* Allergy to gadolinium.
* Type 1 diabetes mellitus or Type 2 diabetes mellitus actively receiving treatment.
* Cognitive impairment that precludes a patient from acting as his or her own agent to provide informed consent.
* Concurrent use of Bosentan.
* Any major medical illnesses or psychiatric impairments that in the treating physician's opinion will prevent administration or completion of protocol therapy ( which may include patients who are elderly, debilitated, or malnourished persons and/or those with renal, hepatic or adrenal insufficiency).
* Pregnant or breast feeding women due potential damage to the fetus
* Inability to undergo MRI or SRS (e.g. due to safety reasons such as presence of a pacemaker).
* Deemed by the treating physician to be unable to eat regular meals.
* Patients currently on beta blockers.
* Patients with a known diagnosis of ongoing alcoholism/alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham (UAB) Department of Radiation Oncology, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Portion: Step 1: Patients with brain metastases requiring SRS and not taking corticosteroids 5 days prior to SRS. Treatment planning MRI may be done within 21 days prior to SRS treatment.
  Step 2: Take Glyburide 1.25mg (twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education- begin glucose monitoring (4 times a day).
  Step 3: 1 week after SRS, return to clinic to review glucose logs- continue glyburide and blood glucose monitoring.
  Step 4: 1 month after SRS, discontinue both glyburide and blood glucose monitoring, undergo MRI.
  Step 5: 3 months after SRS, undergo MRI.
  Glyburide: 1.25mg, twice a day
- Randomized Portion: Step 1: Patients with brain metastases requiring SRS and not taking corticosteroids 5 days prior to SRS.Treatment planning MRI may be done within 21 days prior to SRS treatment.
  Step 2: Randomization (1:1)
  * Group 1: take Glyburide (1.25mg, twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education. Begin glucose monitoring (once a day) {This portion will be double blinded}.
  * Group 2: Take Placebo (1 pill, twice a day by mouth) beginning 5 days prior to SRS. Receive glucose monitoring materials and blood glucose education. Begin glucose monitoring (once a day) {This portion will be double blinded}.
  Step 3: 1 week after SRS, return to clinic to review glucose logs, continue investigation medication, but discontinue glucose monitoring.
  Step 4: 1 month after SRS, discontinue investigation medication, undergo MRI.
  Step 5: 3 months after SRS, undergo MRI.
  Glyburide: 1.25mg, twice a day
  Placebo: 1.25mg, twice a day
Period: Overall Study
Arm/Group | Pilot Portion | Randomized Portion
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: terminated early
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Portion | Randomized Portion | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (0) |  | 41 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Assessed between the time of glyburide initiation and the time of the one month follow-up MRI.
Time Frame: 4 months
Population: Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Primary Outcome: Randomized Portion: Occurrence of Edema Increase and Initiation of Dexamethasone (or Any Corticosteroid Administration With the Purpose of Treating Cerebral Edema)
Description: Assessed between the time of SRS and the time of the one month follow-up MRI.
Time Frame: 4 months
Population: Patients
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Administered Dexamethasone (or Any Corticosteroid Administration With the Purpose of Treating Cerebral Edema)
Description: Measured between the time of SRS and the time of the one and three month post SRS MRI scans.
Time Frame: 4 months
Population: Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With CTCAE Version 4.0 Reportable Toxicities of Grades 2-5.
Description: Incidence of CTCAE version 4.0 reportable toxicities of grades 2-5.
Time Frame: 4 months
Population: Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With CTCAE Version 4.0 Reportable Toxicities of Grades 1-2 Cardiac Disorders or Hepatobiliary Disorders.
Description: Incidence of CTCAE version 4.0 reportable toxicities of grades 1-2 Cardiac Disorders or Hepatobiliary Disorders.
Time Frame: Up to 4 months
Population: no patients were accrued to the randomized portion
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Cerebral Edema Increase as Measured on FLAIR Volumetric Imaging
Description: Defined from MRI taken at the time of SRS and the time of the one and three month post SRS MRI scans.
Time Frame: 4 months
Population: no patients accrued to the randomized portion
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Absolute Volume Change of Index Tumor(s)
Description: Absolute volume change of index tumor(s) that received radiosurgery as manually contoured by the radiation oncologist defined from T1 post gadolinium sequences at the time of SRS and the time of the one and three month post SRS MRI scans.
Time Frame: 4 months
Population: no patients accrued to the randomized portion
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Portion | Randomized Portion
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: While one patient was enrolled, this patient did not experience any AEs.
Arm/Group | Pilot Portion | Randomized Portion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02460874/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT02460874/ICF_001.pdf